CLINICAL TRIAL: NCT02575300
Title: Phase II Study of Ibrutinib in Advanced Carcinoid and Pancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18141
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Carcinoid Tumors; Pancreatic NET
Keywords: neuroendocrine tumors (NETs); gastroenteropancreatic NETs; pancreatic NETs; gastrointestinal (GI) tract NET; advanced carcinoid tumors
MeSH Terms: conditions — Carcinoid Tumor; Adenoma, Islet Cell; Neuroendocrine Tumors | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ibrutinib Therapy (Experimental): Ibrutinib Initial Dose 560 mg by mouth (PO) every day (QD)
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be administered orally once daily and each cycle will be defined as 4 weeks duration. Study treatment should begin within 14 days following enrollment into the study and continue until disease progression, unacceptable toxicity, or withdrawal of consent.
  Other Names: IMBRUVICA®

SUMMARY:
This is a prospective phase II open-label trial, stratifying patients equally into two cohorts consisting of carcinoid tumors and pancreatic neuroendocrine tumors (pNETs). The purpose of this study is to test any good and bad effects of the study drug called Ibrutinib.

The study population will consist of adult patients with histologically confirmed low to intermediate grade NETs of the GI tract, lungs and unknown primary (carcinoid tumors) or pNETs. All patients must be confirmed to have advanced disease. The study will enroll up to 51 patients in two cohorts (30 carcinoid and 21 pNET patients).

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic carcinoid or pancreatic neuroendocrine tumors (pNETs)
* Measureable disease by Response Evaluation Criteria in Solid Tumors (RECIST)
* Tumors must be histologically or cytologically proven and considered low or intermediate grade. Patients with high grade neuroendocrine carcinomas or small cell carcinomas are excluded from the study.
* Evidence of progressive disease within 12 months of study entry
* Allowed prior therapies include: a) Surgery (major surgery at least more than four weeks prior to baseline assessment); b) Locoregional therapy such as: chemoembolization, radio-embolization, radiofrequency ablation, radiotherapy as long as there is progressive measurable disease outside the area of locoregional therapy or there is progression in the previously treated areas; c) Any number of previous lines of systemic therapy. Last treatment before enrollment must have occurred more than 4 weeks for chemotherapy, 6 weeks for antibodies or more than 5 half-lives of prior tyrosine kinase inhibitors (TKIs) or small molecules.
* Prior or concurrent therapy with somatostatin analogs is permitted for patients with secretory NET
* All patients with gastroenteropancreatic NETs must have progressed on (or are intolerant of) prior somatostatin analog.
* Patients with pancreatic NETs must have progressed on (or are intolerant of) either everolimus or sunitinib.
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy 12 weeks or more
* Adequate bone marrow function as shown by: absolute neutrophil count ≥ 1,000/mm^3, Platelets ≥ 100,000/mm^3, Hb > 10 g/dl
* Adequate liver function as shown by: serum bilirubin ≤ 1.5 x ULN, and serum transaminases activity ≤ 2.5 x ULN, with the exception of serum transaminases (< 3 x ULN) if the patient has liver metastases
* Adequate renal function as shown by serum creatinine ≤ 2 mg/dl
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of the administration of the first study treatment. Women must not be lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study.
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.

Exclusion Criteria:

* High grade NET or small cell neuroendocrine carcinoma
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Known positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class III or IV cardiac disease as defined by the New York Heart Association (NYHA) functional classification
* Requirement for anticoagulation with warfarin or similar vitamin K antagonists.
* Requirement for treatment with a strong cytochrome P450 (CYP) 3A4/5
* Prior antitumor therapy within 2 weeks of enrollment (with the exception of somatostatin analogs)
* No other active malignancy within 3 years of enrolment except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least three years
* Any medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib
* Known hypersensitivity to ibrutinib or any component of the ibrutinib formulation
* History of noncompliance to medical regimens or unwillingness to comply with the protocol
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibrutinib Therapy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib Therapy
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Radiographic Response Rate (ORR)
Description: Response rate as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. For this study, measurable disease is defined as the presence of at least one measurable lesion.
  Measurable lesions must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of: 10 mm by CT scan (CT scan slice thickness no greater than 5 mm (when CT scans have slice thickness >5 mm, the minimum size should be twice the slice thickness); 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable); 20 mm by chest X-ray.
  Complete Response (CR): complete disappearance of all target lesions, confirmed by repeat assessments at no less than 4 weeks after the criteria for response are first met. Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Up to 18 months
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib Therapy
Number analyzed (Participants) | 20
Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival at one year. PFS, determined as the time from administration of the initial dose of ibrutinib until objective tumor progression using RECIST, or death. Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib Therapy
Number analyzed (Participants) | 20
months | 3.0 [2.8 to 5.8]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival determined from the time of drug administration to death from any cause.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib Therapy
Number analyzed (Participants) | 20
months | 24.1 [16.5 to NA] — The high end of the range was not reached at time of analysis.

4. Secondary Outcome: Occurrence of Possibly Related Adverse Events (AEs)
Description: Adverse events possibly related to study treatment with Ibrutinib. Safety and tolerability will be assessed according to the NIH/NCI Common TerminologyCriteria for Adverse Events version 4 (CTCAE v4).
Time Frame: Up to 18 months
Population: All participants who received at least one dose of study drug and had at least one adverse event that was possibly probably or definitely related to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib Therapy
Number analyzed (Participants) | 20
Participants | 19

5. Secondary Outcome: Duration of Response
Description: Duration of response, defined as time from first observation of an objective response which is subsequently confirmed, to first disease progression or death due to any cause.
Time Frame: Up to 18 months
Population: No participants experienced objective response
Arm/Group | Ibrutinib Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years, 5 months
Description: SAEs are reported that occurred after first dose of study drug through 30 days after discontinuation of study drug.
Arm/Group | Ibrutinib Therapy
All-Cause Mortality (participants affected / at risk) | 9/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib Therapy (N=20)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib Therapy (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (5)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cataracts (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (17)
Bloating (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 11 (28)
Dyspepsia (Gastrointestinal disorders) | 3 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (9)
Gastrointestinal disorders, other (Gastrointestinal disorders) | 1 (1) — Upset stomach
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorders, other (Gastrointestinal disorders) | 1 (1) — Malabsorption
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (26)
Oral pain (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (13)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (17)
Flu like symptoms (General disorders) | 2 (3)
Irritability (General disorders) | 2 (2)
Neck edema (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (9)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (8)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Memory impairment (Nervous system disorders) | 1 (1)
Parasethesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders-other (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Flushing (Vascular disorders) | 3 (4)
Hot flashes (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 4 (8)
Hypotension (Vascular disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Night sweats
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Sweats (per diary)
General disorders and administration site conditions - Other (General disorders) | 1 (1) — Flu like symptoms
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) — Right ankle sprain
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) — Diabetes
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (5) — Hip pain
Musculoskeletal and connective tissue disorder - other (Musculoskeletal and connective tissue disorders) | 1 (1) — Left hip pain
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Leg muscle cramps
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Basal cell carcinoma
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Brittle nails
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Non-puritic rash
Skin and Subcutaneous tissue disorders -Other (Skin and subcutaneous tissue disorders) | 1 (1) — Hair breakage
Skin and Subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) — Right forearm skin lesion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT02575300/Prot_SAP_000.pdf